CLINICAL TRIAL: NCT02759094
Title: Evaluation of Safety and Effectiveness of the RefluxStop Device in the Management of Gastroesophageal Reflux Disease (GERD)
Brief Title: Evaluation of Safety and Effectiveness of the RefluxStop Device in the Management of GERD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Implantica CE Reflux Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RXI 001
Record Dates: First submitted 2016-04-15; First posted 2016-05-03 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2022-04

CONDITIONS: GERD
Keywords: GERD; Implantable medical device; RefluxStop; Reflux; Gastroesophageal Reflux; Laparoscopy; pH-Monitoring; PPI proton pump inhibitors
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with RefluxStop device (Experimental): All enrolled subjects will receive treatment for their GERD using the RefluxStop device intervention
  Interventions: Device: Treatment with RefluxStop

INTERVENTIONS:
Device: Treatment with RefluxStop — A standard laparoscopic approach will be used to reposition the lower oesophageal sphincter (LES) to its intra-abdominal position. The RefluxStop device will be then positioned and fixed in the gastric funds to ensure intra-abdominal positioning of the GEJ (Gastro-oesophageal Junction) at all time. After confirming proper placement, the laparoscopic implant procedure will be completed and access points will be closed.

SUMMARY:
Prospective, open-label, multi-centre, single arm treatment only trial to evaluate the safety and effectiveness of RefluxStop for the treatment of GERD.

The used medical device "RefluxStop" is an implantable single use sterile device to ensure maintenance of gastro oesophageal junction (GEJ) in an intra-abdominal position to reduce or eliminate GERD.

DETAILED DESCRIPTION:
The study plan will include a screening/baseline visit, a surgical procedure phase with hospital stay until discharge, and study visits at 6 weeks, 3 months and 6 months after device implantation.

A follow-up will be performed annually from years 1-5 to evaluate long-term safety and performance with the intention to collect post-market long-term data using the GERD-HRQL score as a screening tool. Data of subjects who agreed to participate in the long-term safety and performance will be analysed after 1, 2, 3, 4 and 5 years.

At the screening/baseline visit, after signing the informed consent, the eligibility of subjects to receive treatment with the study device will be determined. Eligible subjects will then undergo the device implant procedure.

A standard laparoscopic approach will be used to reposition the lower esophageal sphincter (LES) to its intra-abdominal position. The RefluxStop™ device will then be positioned and fixed in the gastric fundus to ensure intra-abdominal positioning of the GEJ at all time. After confirming proper placement, the laparoscopic implant procedure will be completed and access points will be closed. The procedure will be recorded and saved only with study identification number and without subject ID information. The same applies for images on contrast swallow controlling the device.

Evaluations will be performed daily during hospitalisation and in an additional 3 study visits in the outpatient setting at 6 weeks, 3 months and 6 months. Subjects who have given their consent to participate in the long-term safety and performance follow-up part of the study will be followed annually from year 1-5.

A pathologically low pH in the lower esophagus is correlated to the development of precancerous changes/ Barrett's esophagus and fulminant cancer, as shown in the literature. Barrett's esophagus occurs in 1-2% of the total population while daily acid reflux patients have an incidence of 10-20% depending on the severity of the acid reflux [Modiano, Gerson 2007; Cossentino, Wong 2003]. As many as 48,000 people p.a. die in Europe and the US alone of esophageal adenocarcinoma, the primary cause of which is acid reflux. Therefore, in order to determine whether treatment is maintained in the longer-term, an additional 24-hour pH monitoring and simplified contrast swallow x-ray to verify the position of the device will be performed at 5 years for the benefit of the patients.

These long-term results have also been requested by the U.S. FDA. A quality control of the placement of the device will be categorized for subjects at after surgery, 6 months and 5 year follow-up and at therapy failure.

The position of the device is of utmost importance and will be categorized in the case of therapy failure.

To ensure a proper quality control, the contrast swallow x-ray determining eventual hiatal hernia performed before surgery is repeated at hospital stay after surgery and during the 6-month surgical outcome control and at 5-year follow-up. This x-ray is also used for categorizing the position of the device in a four-graded scale if therapy failure occurs and should be performed by the radiologist using the standard of care post-op contrast swallow.

ELIGIBILITY:
Inclusion Criteria:

* Subject's age >= 18 years and <= 75 years
* Subject is able to undergo general anaesthesia and is a suitable laparoscopic surgical candidate
* Subject is willing and able to participate
* Subject has provided written informed consent after being informed of the study procedure and risks prior to any study-related events
* Subject has documented typical GERD symptoms present for > 6 months which respond to PPIs as anti-GERD medication. Typical symptom of GERD is defined as heartburn, which is a burning epigastric or substernal pain
* Subject requires daily PPI anti GERD medication
* Subject has a 24-hour pH monitoring proven GERD performed taken off any anti reflux medication or after discontinuation for at least 7 days prior to testing. Total distal esophageal pH must be <= 4 for >= 4.5% if time during a 24-hour monitoring

Exclusion Criteria:

* Subject is currently participating in another study involving investigational drugs or devices
* Subject has a history of gastro esophageal surgery, anti-reflux or bariatric procedure
* Subject has a history of endoscopic anti-reflux intervention
* Subject has a history or a suspicion of esophageal or gastric cancer
* Subject has a history of major psychiatric disorder
* Presence of a para-esophageal hernia or sliding hernia of > 3cm determined on endoscopy
* Presence of an esophagitis grade C or D according to the Los Angeles classification
* Presence of esophageal dysmotility disorder such as but not limited to scleroderma, achalasia, Nutcracker oesophagus
* Presence of esophageal stricture or stenosis
* Presence of delayed gastric emptying
* Presence of esophageal or gastric varies
* Subject has a body mass index (BMI) > 35kg/m2
* Female subjects who are pregnant or nursing
* Known sensitivity or allergies to silicone materials
* Subjects who are unable to comply with the protocol requirements
* Subjects with limited life expectancy (< 3 years)
* Intra-operative findings that may preclude conduct of the study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint | at 6 months
  Assessment of incidence of serious adverse device effects (SADEs) and procedure-related serious adverse events (SAEs)
Primary efficacy endpoint | at 6 months
  Percent reduction from baseline of GERD symptoms based on the GERD-HRQL score (questions 1-10). The data will also be presented as the number of subjects obtaining a 50% improvement of the baseline figures, with success defined as 60% of the subjects to reach such score improvement. Thus, the aim of this analysis is to show that the lower limit of the confidence interval exceeds 60%.

SECONDARY OUTCOMES:
Secondary safety endpoint | at 6 weeks, 3 months, 6 months (ADEs and AEs only) and annually years 1-5
  Assessment of incidence of serious adverse device effects (SADEs) and procedure-related serious adverse events (SAEs). Incidence of adverse device effects (ADEs) and procedure-related adverse events (AEs)
Secondary efficacy endpoint: HRQL all other timepoints | measured at baseline, 6 weeks, 3 months and follow-up years 1-5
  Percent reduction from baseline of GERD symptoms based on the GERD-HRQL score (questions 1-10)
Secondary efficacy endpoint: additional questions | measured at baseline, 6 weeks, 3 months, 6 months and follow up years 1-5
  Reduction from baseline of GERD symptoms based on the total GERD-HRQL score (questions 1-10) and individual symptom questions
Secondary efficacy endpoint: 24-hr pH monitoring | measured at baseline, 6 months, 5 years and if therapy failure
  Reduction or normalisation from baseline of the total acid (pH<4) exposure time on 24-hour pH monitoring
Secondary efficacy endpoint: PPI usage | measured at baseline, 6 weeks, 3 months, 6 months and follow up years 1-5
  Reduction from baseline of the percentage of subjects with regular daily PPI usage
Secondary efficacy endpoint: Foregut | measured at baseline, 6 weeks, 3 months, 6 months and follow up years 1-5
  Reduction from baseline of individual foregut questionnaire scores focusing on regurgitation and additional information on dysphagia and odynophagia reported as AEs, or alternatively GERD-HRQL questions >2 and/or >3
Secondary efficacy endpoint: Endoscopy | measured at baseline, 6 months and if therapy failure
  Improvement in esophagitis on upper endoscopy
Secondary efficacy endpoint: device location | measured at hospital stay, 6 weeks, 6 months, 5 years and if therapy failure
  Location and function of the device evaluated by a simplified contrast swallow x-ray with overview pictures of device and LES position during swallowing

OTHER OUTCOMES:
Secondary efficacy subgroup endpoint | per patient any point in the study triggered either by regular daily PPI usage or a GERD-HRQL score with less than 50% improvement compared to baseline, and having been verified as therapy failure via 24-hr pH monitoring and x-ray results
  Reduction or change comparison based on the following subgroups: age, gender, weight and result of baseline total GERD-HRQL score, comparing the following secondary endpoints: the total acid (pH<4) exposure time on routine 24-hour pH monitoring at month 6 and the number and percentage of subjects having verified therapy failure
Exploratory endpoint: procedure complications | during procedure
  Assess any procedure-related complications
Exploratory endpoint: Procedure time | during procedure
  Assess time to perform the procedure
Exploratory endpoint: length of hospital stay | from date of admission to date of discharge, assessed up to 100 months
  Assess length of the subject's hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: László Harsányi, Prof., Principal Investigator — Semmelweis University
Locations (4):
- Hungary (3):
  - Semmelweis University, Budapest
  - University of Debrecen, Kenezy Gyula Teaching Hospital, General Surgery Department, Debrecen
  - Fejer County Szent Gyorgy University Teaching Hospital, Surgical Department, Székesfehérvár
- Clinical Center of Serbia, Clinic for Digestive Surgery, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjelovic M, Harsanyi L, Altorjay A, Kincses Z, Forsell P; Investigators of the RefluxStop Clinical Investigation Study Group. Non-active implantable device treating acid reflux with a new dynamic treatment approach: 1-year results : RefluxStop device; a new method in acid reflux surgery obtaining CE mark. BMC Surg. 2020 Jul 20;20(1):159. doi: 10.1186/s12893-020-00794-9. PMID 32689979